CLINICAL TRIAL: NCT05696873
Title: CoPing strategIes-psyChological flexibiliTy in Patients Hospitalized for Ischemic cardiovascUlaR disEase (PICTURE)
Acronym: PICTURE
Status: Recruiting | Type: Observational
Sponsor: Cardiocentro Ticino (Other)
Responsible Party: Principal Investigator, Marco Valgimigli, Deputy Chief, Cardiocentro Ticino
Other Study IDs: 02_PICTURE
Record Dates: First submitted 2022-12-21; First posted 2023-01-25 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Ischemic Cardiovascular Disease
Keywords: ischemic cardiovascular disease; mental stress; coping strategies; patient's decision to partecipate to clinical trial; adherence to the medications; psychological flexibility; acceptance and commitment therapy; hexaflex; Brief Cope test; MPFI test; CFQ test; MAAS-8 test; CVD-AAQ test
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this trial is to investigate the coping strategies/physiological flexibility construct in patients hospitalized for ischemic cardiovascular disease and the possible association with recurrence of clinical events (any hospitalization and type thereof, myocardial infarction, stroke and death) during the follow up, the patient's decision to participate to clinical trials approved in the center and the adherence to cardiovascular medications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Able to provide informed consent
* Able to speak and read in the local language spoken in hospital
* Admission to the hospital for ischemic cardiovascular disease

Exclusion Criteria:

* Cannot provide written informed consent
* Under judicial protection, tutorship or curatorship
* Unable to understand and follow study-related instructions or unable to comply with study protocol
* Cognitive impairment
* Severe psychiatric disorders according to DSM-5-TR criteria diagnosed in the last 6 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with age ≥ 18 years old and admission to the hospital for ischemic cardiovascular disease.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
coping strategies and the recurrence of any hospitalization and type thereof, myocardial infarction, stroke and death during the follow up period (2 years±14 days from index hospitalization) | 2 years (±14 days) from index hospitalization
  coping strategies (evaluated using Brief COPE test) and the recurrence of clinical events (any hospitalization and type thereof, myocardial infarction, stroke and death) during the follow up period (2 years±14 days from index hospitalization)
psychological flexibility and the recurrence any hospitalization and type thereof, myocardial infarction, stroke and death during the follow up period (2 years±14 days from index hospitalization) | 2 years (±14 days) from index hospitalization
  psychological flexibility construct (evaluated using MPFI test - Multidimensional Psychological Flexibility Inventory test and CFQ test - Cognitive Fusion Questionnaire) and the recurrence of clinical events (any hospitalization and type thereof, myocardial infarction, stroke and death) during the follow up period (2 years±14 days from index hospitalization)
coping strategies and the patient's decision to participate to the clinical trials approved in the centres | at discharge of index hospitalization (up to 4 weeks)
  coping strategies (evaluated using Brief COPE test) and the patient's decision to participate to the clinical trials approved in the centres
psychological flexibility and the patient's decision to participate to the clinical trials approved in the centres | at discharge of index hospitalization (up to 4 weeks)
  psychological flexibility construct (evaluated using MPFI test - Multidimensional Psychological Flexibility Inventory test and CFQ test - Cognitive Fusion Questionnaire) and the patient's decision to participate to the clinical trials approved in the centres
coping strategies and the adherence to cardiovascular medications | 2 years (±14 days) from index hospitalization
  coping strategies (evaluated using Brief COPE test) and the adherence to cardiovascular medications
psychological flexibility and the adherence to cardiovascular medications | 2 years (±14 days) from index hospitalization
  psychological flexibility construct (evaluated using MPFI test and - Multidimensional Psychological Flexibility Inventory test and CFQ test - Cognitive Fusion Questionnaire) and the adherence to cardiovascular medications

SECONDARY OUTCOMES:
each coping strategy and the recurrence of any hospitalization and type thereof, myocardial infarction, stroke and death | 2 years (±14 days) from index hospitalization
  each coping strategy (evaluated using Brief COPE test) and the recurrence of clinical events type (any hospitalization and type thereof, myocardial infarction, stroke and death)
each component of psychological flexibility model and the recurrence of any hospitalization and type thereof, myocardial infarction, stroke and death | 2 years (±14 days) from index hospitalization
  each component of psychological flexibility model (evaluated using MPFI test - Multidimensional Psychological Flexibility Inventory test and CFQ test - Cognitive Fusion Questionnaire) and the recurrence of clinical events type (any hospitalization and type thereof, myocardial infarction, stroke and death)
each coping strategy (evaluated using Brief COPE test) and the participation to each proposed clinical trial, with a particular focus on the SOS-AMI trial | at discharge of index hospitalization (up to 4 weeks)
  each coping strategy (evaluated using Brief COPE test) and the participation to each proposed clinical trial, with a particular focus on the SOS-AMI trial, since it requires copying with the patient decision to self-administer treatment unlike other studies in which treatment is physician-directed
each component of psychological flexibility and the participation to each proposed clinical trial, with a particular focus on the SOS-AMI trial | at discharge of index hospitalization (up to 4 weeks)
  each component of psychological flexibility construct (evaluated using MPFI test and - Multidimensional Psychological Flexibility Inventory test and CFQ test - Cognitive Fusion Questionnaire) and the participation to each proposed clinical trial, with a particular focus on the SOS-AMI trial, since it requires copying with the patient decision to self-administer treatment unlike other studies in which treatment is physician-directed
cognitive fusion and recurrence of cardiovascular events | at 2 years (±14 days) from index hospitalization
  cognitive fusion (evaluated using CFQ test - Cognitive Fusion Questionnaire) and recurrence of cardiovascular events
cognitive fusion and participation to the trials | at discharge of index hospitalization (up to 4 weeks)
  cognitive fusion (evaluated using CFQ test - Cognitive Fusion Questionnaire) and participation to the trials
cognitive fusion and adherence to cardiovascular medications | at 2 years (±14 days) from index hospitalization
  cognitive fusion (evaluated using CFQ test - Cognitive Fusion Questionnaire) and adherence to cardiovascular medications
psychological flexibility evaluated with CVD-AAQ test and cardiovascular events | at 2 years (±14 days) from index hospitalization
  psychological flexibility evaluated with CVD-AAQ test (Cardiovascular Disease Acceptance and Action Questionnaire) and cardiovascular events
psychological flexibility evaluated with CVD-AAQ test and participation to the trials | at discharge of index hospitalization (up to 4 weeks)
  psychological flexibility evaluated with CVD-AAQ test (Cardiovascular Disease Acceptance and Action Questionnaire) and participation to the trials
psychological flexibility evaluated with CVD-AAQ test and adherence to cardiovascular medications | at 2 years (±14 days) from index hospitalization
  psychological flexibility evaluated with CVD-AAQ test (Cardiovascular Disease Acceptance and Action Questionnaire) and adherence to cardiovascular medications

CONTACTS AND LOCATIONS:
Overall Officials: Marco Valgimigli, M.D., Ph.D, Principal Investigator — Cardiocentro Ticino Institute, Ente Ospedaliero Cantonale, Lugano,
Locations (1):
- Enrico Frigoli, Lugano, Switzerland